CLINICAL TRIAL: NCT03209258
Title: An Investigator Initiated and Conducted, International, Multicenter, Stepped Wedge Cluster Randomized Study of a Care Bundle of Physiological Control Strategies in Acute Intracerebral Hemorrhage
Brief Title: The Third, Intensive Care Bundle With Blood Pressure Reduction in Acute Cerebral Hemorrhage Trial
Acronym: INTERACT3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: West China Hospital (Other); Sichuan Credit Pharmaceutical Co., Ltd. (Industry); Takeda (Industry); National Institute for Health Research, United Kingdom (Other Government); Department for International Development, United Kingdom (Other Government); UK Research and Innovation (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Craig Anderson, Executive Director, The George Institute for Global Health, China
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ICH-WCH&GI
Record Dates: First submitted 2017-07-01; First posted 2017-07-06 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Hemorrhage; Stroke; Hypertension; Diabetes; Anticoagulant-induced Bleeding; Cerebral Vascular Disorder; Brain Disorder; Hemorrhage; Intracranial Hemorrhages; Cardiovascular Diseases; Central Nervous System Diseases
Keywords: Stroke; Intracerebral Hemorrhage; Care Bundle; Clinical Trial; Stepped-wedge Cluster; Management; Blood Pressure
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hypertension; Diabetes Mellitus; Cerebrovascular Disorders; Brain Diseases; Hemorrhage; Intracranial Hemorrhages; Cardiovascular Diseases; Central Nervous System Diseases | interventions — Anticoagulation Reversal

STUDY DESIGN:
Intervention Model Description: Stepped-wedge Cluster Randomised Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed care bundle (Other): Management policy to receive a goal-directed care bundle that involves the rapid correction (<1 hour) of physiological variables as soon as the abnormality is recognised and for the control to be maintained in patients for 7 days or hospital discharge (or death, if sooner)
  Interventions: Other: Care bundle of active management
- Usual care group (Other): Patients receive the usual management based on local guidelines and hospital's individual policy.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Care bundle of active management — 1. Intensive BP lowering to systolic target of <140mmHg;
  2. Glucose control target 6.1-7.8 mmol/l for non-diabetic; 7.8-10.0 mmol/l for diabetic patients;
  3. Treatment of pyrexia to a target body temperature ≤37.5 ℃;
  4. Reversal of anticoagulation to target INR <1.5 involving use of vitamin K and prothrombin complex concentrate (PCC) or alternatively, fresh frozen plasma (FFP).
  As the trial is an assessment of care bundle of physiological management, there is some flexibility in the use of particular BP lowering agents and antipyretic agents to achieve targets.
  Other Names: Early intensive BP lowing; Intensive glucose control; Early treatment of pyrexia; Reversal of anticoagulation
  Arms: Goal-directed care bundle
Other: Usual care — Usual care decisions about the location of care delivery, investigations, monitoring, and all treatments will be made by the treating clinical team.
  Arms: Usual care group

SUMMARY:
Continued uncertainty exists over benefits of early intensive blood pressure (BP) lowering in acute intracerebral hemorrhage (ICH), related to the non-significant primary outcomes, patient selection, and discordant results of INTERACT2 and ATACH-II. We designed INTERACT3 to determine the effectiveness of a goal-directed care bundle of active management (intensive BP lowering, glycemic control, treatment of pyrexia and reversal of anticoagulation) vs. usual care in ICH.

INTERACT3 is a large-scale pragmatic clinical trial to provide reliable evidence over the effectiveness of a widely applicable goal-directed care bundle in acute ICH.

DETAILED DESCRIPTION:
Objectives: To determine the effectiveness of a goal-directed care bundle of active management involving early physiological control (intensive blood pressure [BP] lowering, glycemic control, early treatment of pyrexia, and rapid reversal of anticoagulation), versus usual standard of care, on functional outcome (defined by a shift in scores on the modified Rankin scale [mRS] in patients with acute spontaneous intracerebral hemorrhage (ICH).

Study design: An international, multicentre, stepped wedge, cluster randomized clinical trial design involves implementation of a guideline-recommended intervention package applied to patients with ICH as part of routine care. Patients are only excluded if they refuse to have details of their management included and/or participate in the follow-up procedures.

Study site inclusion criteria: Organized systems of acute stroke care; no established comprehensive protocols for the management of patients with ICH; suitable location, infrastructure and willingness to participate in clinical research; large volume of ICH patients (approx. 100 per year). The hospitals will have training, prior to their activation and commencement of the intervention. Data collection at baseline,Day 1, discharge/ Day 7, and 6-month (end of follow-up), will be captured through a web database. Randomized allocation of intervention will be assigned by a statistician not otherwise involved in the study according to a statistical program stratified by the country of the site.

Process Evaluation: Mixed methods were used to explore how the care bundle, a complex intervention, is implemented, as well as to understand clinicians' perspectives, a prospective process evaluation will be conducted alongside the trial implementation. Intervention fidelity, reach, dose, adaption, feasibility and appropriateness of the goal-directed care bundle will be evaluated within the trial.

Economic Evaluation: A multi-country within-trial economic evaluation will be conducted, from each healthcare system's perspective. Healthcare utilisation costs incurred within the initial hospital visit will be estimated using administratively collected hospital records.

Statistical considerations: We anticipate recruiting a minimum of 110 sites in a stepped-wedge design consisting of 3 groups and 4 phases. Each group would therefore include approximately 36-37 sites. We assume an interclass correlation coefficient (ICC) of 0.044 between sites which is similar to that found in the INTERACT2 and recently completed Head Position in Acute Stroke Trial (HeadPoST) trials across Chinese sites. To demonstrate a treatment effect with 90% power and a 2-sided type-I error rate of 5%, each site would need to recruit an average of 18 patients per phase for a total sample size of 7,920 patients. Assuming that 5% of patients will have a missing outcome, each site would need to target an average of 19 patients per phase per site for a total sample size of 8,360 patients. To allow for variability in the number of patients recruited at each site, with very large hospitals expected to recruit up to 50 patients per phase and smaller hospitals recruiting as little as 1 patient per phase in order to allow a broad range of hospitals with variable experience and systems of care for the management of ICH. The sample size would need to be inflated by a factor of approximately 1.3; thus leading to a sample size of up to 25 patients per site per phase (11,000 patients in total). Assuming the worst case scenario for the effect of cluster size variability on power, this sample size would still provide at least 80% power. This sample size provides 90% power to determine a treatment effect of a 5.6% absolute improvement in the proportion of patients experiencing a bad outcome (modified Rankin scale [mRS] scores of 3-6), from 55.6% down to 50%. This also translates to a 10% relative risk reduction (relative risk of 0.90). All analyses will be undertaken at the patient level on an intention-to-treat basis at each center using Generalised Estimating Equations (GEE) or random-effects regression to account for clustering.

Ethics consideration: A mixed consent process is proposed, according to local/national rules and regulations, for the following protocol:

Cluster Guardian consent or appropriate approval (e.g. signed by General Manager or Chief Executive of hospital, or Head of Neurology/Stroke Department) for the goal-directed care bundle to be the new usual management for patients with ICH;

With one of the following:

(i). Individual standard consent for the collection of data through in-person assessment and data extraction from medical records during the hospital stay and follow-up, and for release of personalized information for research purposes to allow centralized follow-up at 6-month after admission, or (ii). Opt-out/withdraw consent for collection of data through in-person assessment and data extraction from medical records during the hospital stay and follow-up, and for release of personalized information for research purposes to allow centralized follow-up at 90 days after admission.

Data management: The internet based data management system is managed at the George Institute for Global Health, which has extensive experience in clinical trial data capture and security. The George Institute has in place system security SOP with VeriSign SSL digital certification and encrypted HTTPS connection. Only staff listed in the delegation log will be given unique individual password to access the internet-based data management system.

Data collection: Paper CRFs will be provided for sites preferring to use these for the initial collection of data. These forms will be used as source document and will need to be signed and dated by the investigator completing the form. All computerized forms will be electronically signed (by use of the unique password) by the authorized study staff and all changes made following the initial entry will have an electronic dated audit trail. It is the requirement that the collection of data and transfer of information for the 90 day follow-up assessment has to be approved by the local IRB for each site.

Collarboration: Central international coordination is from GI, China and together with regional coordinating centers established and located in Sydney, and Santiago, Chile, the study will be overseen by an International Steering Committee comprised of world experts in the fields of stroke, neurocritical care, neurology, geriatrics, cardiovascular epidemiology and clinical trials. The investigators of the 110 participating hospitals will be administratively tied through a structure designed to enhance effective communication, collaboration and study monitoring by maintaining operations through adherence to a common protocol.

Data Safety & Monitoring Board (DSMB): The DSMB will review the safety, ethics and outcomes of the study.The DSMB will be governed by a charter that will outline their responsibilities, procedures and confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Acute stroke syndrome that is due to presumed spontaneous ICH, confirmed by clinical history and a CT scan within 6 hours of stroke onset without/without contrast, and if an CT angiogram is also undertaken as part of routine care.
* Presentation to hospital within 6 hours of stroke onset.

Exclusion Criteria:

* Definite evidence that the ICH is secondary to a structural abnormality in the brain (eg an AVM, intracranial aneurysm, tumour, trauma, or previous cerebral infarction) or previous thrombolysis.
* A high likelihood that the patient will not adhere to the study treatment and follow-up regimen. In each case, the decision about the patient's eligibility will be based on the attending clinician's interpretation of the above eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7067 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Shift ('improvement') in functional recovery (death or disability) defined by the modified Rankin Scale (mRS) | 6 months
  modified Rankin Scale is a measure of physical function at 6 months, analyzed as an ordinal outcome (categories scored as 0 'no symptoms' to 5 as 'fully dependent, and 6 as death)

SECONDARY OUTCOMES:
Shift ('improvement') in survival and neurological impairment defined by scores on the National Institutes of Health Stroke Scale (NIHSS) | 7 days
  measure of physical function
Death or disability defined by scores of 3-6 on the mRS | 6 months
  measure of physical function
Death | 6 months
  measure of vital status
Disability defined by scores 3-5 on the mRS | 6 months
  measure of physical function
Health-related quality of life (HRQoL) | 6 months
  measure of quality of life on the EQ5D scale
Duration of initial hospitalization | 6 months
  measure of severity and service use
Residence | 6 months
  measure of patient living status (e.g. home, high care)

CONTACTS AND LOCATIONS:
Overall Officials: Craig S Anderson, PhD, Principal Investigator — The George Institute for Global Health, China; Chao You, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ren X, Li Q, Ouyang M, Billot L, Chen X, Venturelli PM, de Silva A, Nguyen TH, Wahab KW, Pandian JD, Wasay M, Pontes-Neto OM, Abanto C, Arauz A, You C, Ma L, Hu X, Anderson C, Wang X, Song L; as the INTERACT3 Investigators. Mediation Analysis to Identify Individual Component Effects of the Care Bundle to Improve Functional Outcome After ICH in the INTERACT3 Study. Neurology. 2025 Oct;105(7):e214070. doi: 10.1212/WNL.0000000000214070. Epub 2025 Sep 12. PMID 40939125
- [Derived] Hu X, Ouyang M, Xu J, Liu Y, Li X, Jiang Y, Chen X, Billot L, Li MBiostat Q, Malavera A, Venturelli PMO, de Silva A, Thang NH, Wahab KW, Pandian JD, Wasay M, Pontes-Neto OM, Abanto C, Arauz A, Li Z, Chen M, Wang X, Yang C, Xin X, Jiang D, Zheng J, Yu Z, Xiao A, Tao C, Chen L, Wu B, Li H, Anderson CS, You C, Song L, Ma L; INTERACT3 Investigators. Surgical outcomes from haematoma evacuation for intracerebral haemorrhage in the INTERACT3 study. Lancet Reg Health West Pac. 2025 Aug 28;62:101669. doi: 10.1016/j.lanwpc.2025.101669. eCollection 2025 Sep. PMID 40927652
- [Derived] Wang X, Ren X, Li Q, Ouyang M, Chen C, Delcourt C, Chen X, Wang J, Robinson T, Arima H, Ma L, Hu X, You C, Li G, Jie Y, Lin Y, Billot L, Munoz-Venturelli P, Martins S, Pontes-Neto OM, Liu L, Chalmers J, Carcel C, Song L, Anderson CS; INTERACT Investigators. Effects of blood pressure lowering in relation to time in acute intracerebral haemorrhage: a pooled analysis of the four INTERACT trials. Lancet Neurol. 2025 Jul;24(7):571-579. doi: 10.1016/S1474-4422(25)00160-7. PMID 40541207
- [Derived] Ouyang M, Anjum A, Mc Cawley FG, Wasay M, Ma L, Hu X, Chen X, Malavera A, Li X, Venturelli PM, Silva HA, Thang NH, Wahab KW, Pandian JD, Pontes-Neto OM, Abanto C, Cano-Nigenda V, Arauz A, You C, Jan S, Song L, Anderson CS, Liu H; INTERACT3 Investigators. Implementation of a goal-directed Care Bundle for intracerebral hemorrhage: Results of embedded process evaluation in the INTERACT3 trial. PLOS Glob Public Health. 2024 Dec 19;4(12):e0003711. doi: 10.1371/journal.pgph.0003711. eCollection 2024. PMID 39700102
- [Derived] Ma L, Hu X, Song L, Chen X, Ouyang M, Billot L, Li Q, Malavera A, Li X, Munoz-Venturelli P, de Silva A, Thang NH, Wahab KW, Pandian JD, Wasay M, Pontes-Neto OM, Abanto C, Arauz A, Shi H, Tang G, Zhu S, She X, Liu L, Sakamoto Y, You S, Han Q, Crutzen B, Cheung E, Li Y, Wang X, Chen C, Liu F, Zhao Y, Li H, Liu Y, Jiang Y, Chen L, Wu B, Liu M, Xu J, You C, Anderson CS; INTERACT3 Investigators. The third Intensive Care Bundle with Blood Pressure Reduction in Acute Cerebral Haemorrhage Trial (INTERACT3): an international, stepped wedge cluster randomised controlled trial. Lancet. 2023 Jul 1;402(10395):27-40. doi: 10.1016/S0140-6736(23)00806-1. Epub 2023 May 25. PMID 37245517
- [Derived] Billot L, Song L, Hu X, Ma L, Ouyang M, Chen X, You C, Anderson CS; INTERACT3 Investigators. Statistical Analysis Plan for the INTEnsive Care Bundle with Blood Pressure Reduction in Acute Cerebral Hemorrhage Trial: A Stepped-Wedge Cluster Randomized Controlled Trial. Cerebrovasc Dis. 2023;52(3):251-254. doi: 10.1159/000526384. Epub 2022 Sep 5. PMID 36063792
- [Derived] Ouyang M, Anderson CS, Song L, Malavera A, Jan S, Cheng G, Chu H, Hu X, Ma L, Chen X, You C, Liu H. Process Evaluation of an Implementation Trial: Design, Rationale, and Early Lessons Learnt From an International Cluster Clinical Trial in Intracerebral Hemorrhage. Front Med (Lausanne). 2022 Jun 15;9:813749. doi: 10.3389/fmed.2022.813749. eCollection 2022. PMID 35783649
- [Derived] Song L, Hu X, Ma L, Chen X, Ouyang M, Billot L, Li Q, Munoz-Venturelli P, Abanto C, Pontes-Neto OM, Antonio A, Wasay M, Silva A, Thang NH, Pandian JD, Wahab KW, You C, Anderson CS; INTERACT3 investigators. INTEnsive care bundle with blood pressure reduction in acute cerebral hemorrhage trial (INTERACT3): study protocol for a pragmatic stepped-wedge cluster-randomized controlled trial. Trials. 2021 Dec 20;22(1):943. doi: 10.1186/s13063-021-05881-7. PMID 34930428
- [Derived] Ouyang M, Anderson CS, Song L, Jan S, Sun L, Cheng G, Chu H, Hu X, Ma L, Chen X, You C, Liu H. Implementing a Goal-Directed Care Bundle after Acute Intracerebral Haemorrhage: Process Evaluation for the Third INTEnsive Care Bundle with Blood Pressure Reduction in Acute Cerebral Haemorrhage Trial Study in China. Cerebrovasc Dis. 2022;51(3):373-383. doi: 10.1159/000520669. Epub 2021 Dec 20. PMID 34929690